CLINICAL TRIAL: NCT02284997
Title: The Effect of an Eyelid Warming Device for the Management of Meibomian Gland Dysfunction
Acronym: Hummingbird
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Waterloo (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 20246
Record Dates: First submitted 2014-11-03; First posted 2014-11-06 (Estimated); Last update posted 2015-05-29 (Estimated); Status verified 2015-05

CONDITIONS: Meibomian Gland Dysfunction (MGD)
MeSH Terms: conditions — Meibomian Gland Dysfunction

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Treatment (Experimental): Participants will be instructed to use a warming MGDRx® EyeBag for minimum of 10 minutes, twice a day
  Interventions: Device: MGDRx® EyeBag
- Control (No Intervention): No treatment

INTERVENTIONS:
Device: MGDRx® EyeBag — Class 1 Medical Device, registered with the Medicines and Healthcare products Regulatory Agency. UK Patent: GB2421687B. The EyeBag is made of silk and 100% brushed black cotton and filled with flax / linseed. When heated, this device is intended to warm the eyelids. This melts the meibum and clears the meibum obstruction of the MGs.
  Arms: Treatment

SUMMARY:
Along the edge of the eyelids, there are glands (meibomian glands) that produce and deliver oils (meibum) onto the tear film. These oils serve to slow down the evaporation of tears. The meibomian glands may become obstructed due to change in meibum quality. When meibum thickens and solidifies, it plugs the gland openings and oils can no longer reach the tear film. The blockage of the glands is the primary cause of meibomian gland dysfunction (MGD), and may result in symptoms of dry eye (burning, stinging, grittiness, etc.). The typical treatment for MGD is a procedure called "warm compresses". It is a combination of applying heat and pressure to the eyelids for approximately 10 minutes to melt the meibum, unplug the gland openings, and allow oils to flow normally onto the tear film once again. One way to apply heat to the eyelids is by using the MGDRx® EyeBag. The EyeBag is microwaved for 30-40 seconds under full power, and is placed over the closed eyes for approximately 10 minutes. The eyes are gently massaged afterwards.

The purpose of this study is to determine how effective the EyeBag is at improving MGD and dry eye symptoms.

ELIGIBILITY:
Inclusion Criteria:

A person is eligible for inclusion in the study if he/she:

1. Is at least 17 years of age and has full legal capacity to volunteer;
2. Has read and signed an information consent letter;
3. Is willing and able to follow instructions and maintain the appointment schedule;
4. OSDI score ≥ 23;
5. Meibomian gland score of ≤ 9 (out of 15).
6. Is on a stable dry eye regimen (if applicable) within the past 4 weeks, and is willing to maintain this regimen
7. Agree to using MetricWire for online data entry
8. Is not a contact lens wearer (Infrequent soft contact lens wearer is acceptable (wear contact lenses for maximum 2 days of the week)).

Exclusion Criteria:

A person will be excluded from the study if he/she:

1. Is participating in any concurrent clinical or research study;
2. Has any known hypersensitivity to flax, linseed or any of the other constituents of the EyeBag
3. Has any known active* ocular disease and/or infection;
4. Has a systemic condition that in the opinion of the investigator may affect a study outcome variable;
5. Is using any systemic or topical medications that in the opinion of the investigator may affect a study outcome variable
6. Has known sensitivity to the diagnostic pharmaceuticals to be used in the study;
7. Is pregnant, lactating or planning a pregnancy at the time of enrolment, as determined verbally;
8. Is aphakic;
9. Has undergone refractive error surgery; * For the purposes of this study, active ocular disease is defined as infection or inflammation which requires therapeutic treatment. An exception is made for lid abnormalities (blepharitis, meibomian gland dysfunction, papillae), corneal and conjunctival staining and dry eye. Neovascularization and corneal scars are the result of previous hypoxia, infection or inflammation and are therefore not active.

Min Age: 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2014-11; Primary Completion 2015-04 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
Meibomian gland score (MGS) | Baseline
  Prior to treatment (if applicable). Scale 0-3. 0: no secretion, 1: inspissated (toothpaste), 2: cloudy with debris, 3: clear
Meibomian gland score (MGS) | 8 weeks after baseline/treatment visit
  Eight weeks after treatment (if applicable). Scale 0-3. 0: no secretion, 1: inspissated (toothpaste), 2: cloudy with debris, 3: clear
Meibomian gland yielding liquid secretions (MGYLS) | Baseline
  Prior to treatment (if applicable). MGYLS is the number of glands with MGS grade 2 or higher.
Meibomian gland yielding liquid secretions (MGYLS) | 8 weeks after baseline/treatment visit
  MGYLS is the number of glands with MGS grade 2 or higher.
Ocular Surface Disease Index Score (OSDI) | Baseline
  Prior to treatment (if applicable). The OSDI is a questionnaire that consists of 12 questions about ocular irritation and the effect of dry eye on vision. For every question, participants check a score between 0 and 4, where 0 equals "none of the time" and 4 equals "all of the time". OSDI scores are calculated according to: OSDI = [(sum of scores for all questions answered)*100] / [(total number of questions answered)*4]. The possible range of the OSDI score is 0 to 100.
Ocular Surface Disease Index Score (OSDI) | 8 weeks after baseline/treatment visit
  The OSDI is a questionnaire that consists of 12 questions about ocular irritation and the effect of dry eye on vision. For every question, participants check a score between 0 and 4, where 0 equals "none of the time" and 4 equals "all of the time". OSDI scores are calculated according to: OSDI = [(sum of scores for all questions answered)*100] / [(total number of questions answered)*4]. The possible range of the OSDI score is 0 to 100.

CONTACTS AND LOCATIONS:
Overall Officials: Lyndon Jones, PhD, Principal Investigator — CCLR, University of Waterloo
Locations (1):
- Centre for Contact Lens Research, University of Waterloo, Waterloo, Ontario, Canada